CLINICAL TRIAL: NCT00373490
Title: MK0683 Phase1 Clinical Study - Solid Tumor -
Brief Title: A Study of Oral Suberoylanilide Hydroxamic Acid (Vorinostat) in Patients With Solid Tumors (0683-048)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-048; MK0683-048; 2006_030
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2009-05-20 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — Vorinostat

ARMS (2):
- Vorinostat 600 mg (Experimental): 600 mg daily (300 mg twice daily [b.i.d.]) for 3 consecutive days followed by 4 days of rest.
  Interventions: Drug: Vorinostat
- Vorinostat 400 mg (Experimental): 400 mg once daily (400 mg q.d.) continuous daily dosing for 21 days.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — 600 mg daily (300 mg twice daily [b.i.d.]) for 3 consecutive days followed by 4 days of rest.
  Other Names: MK-0683; Suberoylanilide Hydroxamic Acid (SAHA)
  Arms: Vorinostat 600 mg
Drug: Vorinostat — 400 mg once daily (400 mg q.d.) continuous daily dosing for 21 days.
  Other Names: MK-0683; Suberoylanilide Hydroxamic Acid (SAHA)
  Arms: Vorinostat 400 mg

SUMMARY:
This is a clinical study to evaluate the safety and pharmacokinetics of an overseas determined maximum tolerated dose (MTD) of MK-0683 (vorinostat) in a Japanese patient population with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically diagnosed solid tumor in whom no standard therapy is available or the malignancy is refractory to standard therapy

Exclusion Criteria:

* Patients with history of immunotherapy, radiotherapy, surgery, or chemotherapy during the previous 4 weeks
* Any uncontrolled concomitant illness
* Pregnant or breast-feeding
* Serious drug or food allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Doi T, Hamaguchi T, Shirao K, Chin K, Hatake K, Noguchi K, Otsuki T, Mehta A, Ohtsu A. Evaluation of safety, pharmacokinetics, and efficacy of vorinostat, a histone deacetylase inhibitor, in the treatment of gastrointestinal (GI) cancer in a phase I clinical trial. Int J Clin Oncol. 2013 Feb;18(1):87-95. doi: 10.1007/s10147-011-0348-6. Epub 2012 Jan 11. PMID 22234637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I. First participant started on study therapy on 18-Jul-2006. Study was multicenter (total of 3 sites).
Pre-assignment Details: Study of 2 doses of vorinostat (MK-0683) in participants with solid tumors who failed standard therapy. >= 3 participants were enrolled at each dose. In the case of a dose level toxicity, a maximum of 6 participants were enrolled per level. If no safety problems, a total of 10 participants were evaluated for pharmacokinetics.
Groups:
- Vorinostat 600 mg: 600 mg daily (300 mg twice daily [b.i.d.]) for 3 consecutive days followed by 4 days of rest (repeated 3 times over 21 days)
Period: Overall Study
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Started | 10 | 6
Completed | 1 | 0
Not Completed | 9 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 9 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.4) | 53.3 (12) | 57.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 4 | 12
Prior chemotherapy regimens [Median (Full Range); unit: Number of prior chemotherapy regimens] | 3.5 [2 to 6] | 4.5 [3 to 6] | 4 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: Dose Limiting Toxicity = Drug-related side effects that are serious enough to prevent an increase in dose or level of that treatment
Time Frame: 21 Days (first cycle)
Population: Six (6) participants received vorinostat at 400 mg once daily. Of these, 2 participants did not complete the first cycle resulting in the drug compliance falling below 75%, and thus these participants were excluded from the DLT assessment.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 10 | 4
Participants | 0 | 2

2. Secondary Outcome: Area Under the Curve (AUC(0-infinity)) at Day 1 (600 mg and 400 mg)
Description: Area Under Curve (AUC(0-infinity))=Area under the plasma concentration versus time curve (AUC) from time zero to extrapolated infinite time (o- ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). At 600 mg, t=12 hours and at 400 mg, t=24 hours.
Time Frame: Day 1 (600 mg and 400 mg)
Population: Six (6) participants received vorinostat at 400 mg once daily. Of these, one (1) participant had missing Pharmacokinetics Data on Day 1 because the participant vomited after administration on Day 1.
Measure: Geometric Mean (Standard Deviation); unit: μM·hr
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 10 | 5
μM·hr | 3.94 (1.56) | 7.75 (2.79)

3. Secondary Outcome: Area Under the Curve (AUC(0-infinity)) at Day 3 (600 mg)
Description: Area Under Curve (AUC(0-infinity))=Area under the plasma concentration versus time curve (AUC) from time zero to 24 ｈours. It is obtained from AUC (0 - 12) plus AUC (12 - ∞)
Time Frame: Day 3 (600 mg)
Measure: Geometric Mean (Standard Deviation); unit: μM·hr
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 10 | 0
μM·hr | 4.15 (2.15) |

4. Secondary Outcome: Area Under the Curve (AUC(0-infinity) at Day 21 (400 mg)
Description: Area Under Curve (AUC(0-infinity))=Area under the plasma concentration versus time curve (AUC) from time zero to 24 ｈours. It is obtained from AUC (0 - 24) plus AUC (24 - ∞)
Time Frame: Day 21 (400 mg)
Population: Six (6) participants received vorinostat at 400 mg once daily. Of these, four (4) participants had missing Pharmacokinetics Data on Day 21 because they did not receive study drug on day 21.
Measure: Geometric Mean (Standard Deviation); unit: μM·hr
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 0 | 2
μM·hr |  | 8.3 (0.04)

5. Secondary Outcome: Maximum Concentration (Cmax) at Day 1 (600 mg and 400 mg)
Time Frame: Day 1 (600 mg and 400 mg)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μM
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 10 | 5
μM | 1.17 (0.43) | 1.62 (0.52)

6. Secondary Outcome: Maximum Concentration (Cmax) at Day 3 (600 mg)
Time Frame: Day 3 (600 mg)
Measure: Geometric Mean (Standard Deviation); unit: μM
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 10 | 0
μM | 1.32 (0.75) |

7. Secondary Outcome: Maximum Concentration (Cmax) at Day 21 (400 mg)
Time Frame: Day 21 (400 mg)
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: μM
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Number analyzed (Participants) | 0 | 2
μM |  | 2.04 (0.78)

ADVERSE EVENTS:
Arm/Group | Vorinostat 600 mg | Vorinostat 400 mg
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/6
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 600 mg (N=10) | Vorinostat 400 mg (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 600 mg (N=10) | Vorinostat 400 mg (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
EAR CONGESTION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (5) | 1 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 1 (1)
ACETONAEMIC VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 2 (4)
CONSTIPATION (Gastrointestinal disorders) | 6 (7) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 4 (27) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
ERUCTATION (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 8 (28) | 6 (12)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (2)
VOMITING (Gastrointestinal disorders) | 5 (14) | 5 (13)
CATHETER SITE PAIN (General disorders) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 8 (48) | 4 (5)
FEELING ABNORMAL (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 2 (11) | 0 (0)
OEDEMA (General disorders) | 2 (2) | 3 (3)
PAIN (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 2 (3)
THIRST (General disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME SHORTENED (Investigations) | 1 (2) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4) | 2 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 (12) | 3 (3)
BLOOD ALBUMIN DECREASED (Investigations) | 2 (2) | 3 (4)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (5) | 3 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (12) | 3 (6)
BLOOD CALCIUM DECREASED (Investigations) | 2 (5) | 0 (0)
BLOOD CHLORIDE DECREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 5 (9) | 5 (12)
BLOOD GLUCOSE DECREASED (Investigations) | 3 (4) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 6 (11) | 5 (8)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 2 (2) | 3 (3)
BLOOD MAGNESIUM DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD MAGNESIUM INCREASED (Investigations) | 3 (5) | 3 (6)
BLOOD PHOSPHORUS DECREASED (Investigations) | 5 (11) | 1 (2)
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 (0) | 1 (2)
BLOOD POTASSIUM INCREASED (Investigations) | 3 (12) | 1 (1)
BLOOD SODIUM DECREASED (Investigations) | 4 (6) | 1 (1)
BLOOD URIC ACID DECREASED (Investigations) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 2 (3) | 2 (4)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 5 (6) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 5 (12) | 4 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (7) | 1 (3)
PLATELET COUNT DECREASED (Investigations) | 3 (6) | 6 (14)
PROTEIN TOTAL DECREASED (Investigations) | 0 (0) | 1 (1)
PROTEIN URINE PRESENT (Investigations) | 2 (2) | 2 (4)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 1 (1) | 0 (0)
URINARY SEDIMENT ABNORMAL (Investigations) | 2 (8) | 0 (0)
URINE BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
UROBILIN URINE PRESENT (Investigations) | 1 (6) | 1 (1)
WEIGHT DECREASED (Investigations) | 6 (7) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 (6) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (3) | 1 (1)
WHITE BLOOD CELLS URINE (Investigations) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 9 (45) | 6 (11)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (4) | 1 (2)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 3 (3)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 0 (0) | 1 (2)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (3)
INSOMNIA (Psychiatric disorders) | 1 (4) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NAIL BED INFLAMMATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.